CLINICAL TRIAL: NCT05837221
Title: Role of Human Microbiome in Head and Neck Cancer
Brief Title: Microbiome in Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-0016.cc; P50CA261605 (NIH)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer; Lip Cancer; Oral Cancer; Pharynx Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lip Neoplasms; Mouth Neoplasms; Pharyngeal Neoplasms | interventions — Metabolic Flux Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Oral Squamous Cell Carcinoma Saliva Sample Group: Saliva will be collected at least 30 minutes after subjects stop eating, drinking, chewing gum, and smoking. Subjects will be instructed to spit saliva into a collection tube. The saliva will be split into two aliquots, one that is immediately frozen at
  -80C and one that is mixed 1:1 with pre-reduced tryptic soy broth, L-cysteine, and glycerol then frozen at -80C to preserve the viability of microorganisms.
  Interventions: Diagnostic Test: Metagenomic sequencing; Diagnostic Test: Metabolic analysis
- Non Oral Squamous Cell Carcinoma Saliva Sample Group: Saliva will be collected at least 30 minutes after subjects stop eating, drinking, chewing gum, and smoking. Subjects will be instructed to spit saliva into a collection tube. The saliva will be split into two aliquots, one that is immediately frozen at
  -80C and one that is mixed 1:1 with pre-reduced tryptic soy broth, L-cysteine, and glycerol then frozen at -80C to preserve the viability of microorganisms.
  Interventions: Diagnostic Test: Metagenomic sequencing; Diagnostic Test: Metabolic analysis
- Oral Squamous Cell Carcinoma Stool Sample Group: Stool collection methods may differ depending on the patient. The aim is to collect fresh stool samples, those that are available will be collected during the study visit. If a patient is unable to give a sample at the visit, samples may be collected at home using the OMNIgene-GUT and OMNImet-GUT kits (DNA Genotek, Inc.).
  Interventions: Diagnostic Test: Metagenomic sequencing; Diagnostic Test: Metabolic analysis
- Non Oral Squamous Cell Carcinoma Stool Sample Group: Stool collection methods may differ depending on the patient. The aim is to collect fresh stool samples, those that are available will be collected during the study visit. If a patient is unable to give a sample at the visit, samples may be collected at home using the OMNIgene-GUT and OMNImet-GUT kits (DNA Genotek, Inc.).
  Interventions: Diagnostic Test: Metagenomic sequencing; Diagnostic Test: Metabolic analysis

INTERVENTIONS:
Diagnostic Test: Metagenomic sequencing — Shotgun metagenomic sequencing will characterize cancer-associated changes in microbial functional capacity and species/strain-level taxonomic profiles. Metagenomics will provide data on microbial functional capacity along with broader taxonomic classifications.
Diagnostic Test: Metabolic analysis — Metabolic analysis will be conducted using LC/MS-based metabolic analysis. A targeted approach will quantify a panel of 30 compounds including Trp pathway products while a non-targeted approach, when applied to both lipid and aqueous phase compounds, will profile relative changes in compounds that may influence host

SUMMARY:
This study aims to determine whether dysbiosis actively contributes to HNSCC and if so, the underlying molecular mechanisms.

DETAILED DESCRIPTION:
HNSCCis a lethal cancer with a 5-year survival rate below 50%. Although smoking, alcohol intake, and human papillomavirus (HPV) infection are linked to HNSCC, only a small proportion of individuals exposed to these factors develop cancer and not all cases progress. Thus, additional environmental or host factors must contribute to HNSCC. The Study Team and others have observed significant oral dysbiosis in human HNSCC cases, both before and after treatment. This study aims to determine whether dysbiosis actively contributes to HNSCC and if so, the underlying molecular mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects equal to or above the age of 18.
2. Patients who are seen and evaluated by a provider within the adult Otolaryngology clinic at the University of Colorado Health.
3. Patients that present with a diagnosis of OSCC.
4. An equal number of age-matched patients who are visiting the clinic for reasons other than OSCC diagnoses, as the control group.
5. Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

1. Subjects under the age of 18 or over the age of 100
2. Subjects unwilling to particiapte

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to enroll 60 patients total - 30 with oral squamous cell carcinoma (OSCC) who are treatment naïve, and 30 who are non-OSCC control patients, who will be age matched to their OSCC counterparts. Estimates show that Dr. Goddard's practice sees approximately 3 treatment naïve OSCC cases per month. We estimate that we can enroll 30-40 of these cases and an equal number of controls in the first 18 months of this study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Characterize human dysbiosis | Day 1
  Stool and saliva samples will be collected from participants, allowing us to reproduce human dysbiosis and analyze whether HNSCC affects one's microbiome composition. Metagenomic sequencing will be conducted through use of DNA extraction, library generation and Illumina sequencing. At least 30 million paired-end 2x150bp metagenomic reads will be generated per sample using the Illumina NovaSeq platform.
Characterize human metabolomics | Day 1
  Through our stool and saliva samples we will be able to characterize metagenomic and metabolic signatures in treatment naïve OSCC and non-OSCC patients. Metabolic analysis will be conducted using LC/MS-based metabolic analysis. A targeted approach will quantify a panel of 30 componds including Trp pathway products, while a non-targeted approach, when applied to both lipid and aqueous phase compounds, will profile relative changes in compounds that may influence host and metabolic and immune statuses.
Integrative multi-omic data analysis and biomarker discovery | Day 365
  We expect to find that specific sets of microbial and host factors interact with each other to promote OSCC.

SECONDARY OUTCOMES:
Impact of human dysbiosis on OSCC development in mice | Day 10-Day 100
  Freshly collected saliva and stool samples from 10 subjects of each treatment category will be used to reconstitute microbiota.
Monitor tumor size | Day 10-Day 100
  Tumor size (both weight and size) will be monitored using Bli-imaging. These measures will be assessed between treatment groups by ANOVA or analysis of variance testing.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Long E Lu, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States